CLINICAL TRIAL: NCT01430832
Title: The Long-Term Developmental Outcomes of Extreme Prematurity: Correlations With Maternal Post-Traumatic Symptoms, Parental Stress and Post-Traumatic Growth, 5-15 Years Postpartum
Brief Title: Developmental Outcomes of Extreme Prematurity, 5-15 Years Postpartum
Status: Terminated | Type: Observational
Why Stopped: Recruitment Status
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-10-8121-LG-CTIL
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Preterm Infants; Post Traumatic Stress Disorder; Emotional Stress; Infant, Very Low Birth Weight
Keywords: PTSD; Preterm; Premature; VLBW
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress, Psychological; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Development: The infant's development level will be assessed using a phone interview with parents
- Abnormal Development: The infant's level of development will be assessed using a phone interview with parents

SUMMARY:
The purpose of this study is to assess the emotional well being of mothers to preterm infants with ELBW 5-15 years after the birth. Post-traumatic symptoms and parental stress levels will be taken into consideration. In addition, the correlation between the infant's development and the mother's emotional state will be analyzed.

DETAILED DESCRIPTION:
Medical records of the children will be used for information in four categories: prenatal, birth, development,and demographic information. Parents will be contacted and interviewed regarding the child's development. In addition, they will complete the following questionnaires: PPQ-II Perinatal PTSD Questionnaire- modified, PTGI -The Posttraumatic Growth Inventory,Parental Stress Index- Short Form- PSI-SF, and Life Events questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infant
* Very low birth weight or extremely low birth weight

Exclusion Criteria:

* Missing information regarding birth week and weight

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants are children born at Sheba Medical center between the years 1995-2006.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2011-09-01; Primary Completion 2011-11-01 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Not relevant | Not relevant

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Gabis, MD, Principal Investigator — Sheba Medical Center; Gabi Zerach, Ph.D, Principal Investigator — Ariel University; Shefer Shahar, Ph.D, Study Director — Sheba Medical Center; Adi Elsing, BA, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided